CLINICAL TRIAL: NCT05740371
Title: SAICoDis - Safety of Argatroban Infusion in Conduction Disturbances. A Prospective, Open, Multicenter Safety Study to Investigate Conduction Disturbances in Patients Receiving Argatroban Therapy.
Brief Title: Safety of Argatroban Infusion in Conduction Disturbances
Acronym: SAICoDis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanabe Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARG-E08; 2016-003521-42 (EudraCT Number)
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Stable Coronary Artery Disease (CAD); Unstable Angina (Troponin Negative)
MeSH Terms: conditions — Angina, Unstable | interventions — argatroban

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Argatroban (Other)
  Interventions: Drug: Argatroban

INTERVENTIONS:
Drug: Argatroban — Patients received an intravenous (i.v.) bolus of 300 μg/kg argatroban administered over a span of 3 to 5 minutes followed by the i.v. infusion of argatroban at 20 μg/kg/min until the end of the procedure. ACT was checked 5 minutes after bolus dose.
  If ACT remained below the target of 300 s, the patient received an additional i.v. bolus injection of 150 μg/kg and the infusion dose was raised up to 30 μg/kg/min.
  In cases ACT > 450 s, the infusion was reduced to 15 μg/kg/min and the value was checked again after 5 minutes.
  As soon as the target ACT (between 300 s and 450 s) was reached, infusion dose remained unchanged during the PCI procedure.
  Depending on clinical relevancy further ACT assessments were possible.
  Other Names: Arganova; Argatra; Novastan

SUMMARY:
To determine change of QTc interval during intravenous argatroban infusion in patients undergoing percutaneous coronary intervention (PCI)

DETAILED DESCRIPTION:
Primary objective:

To determine change of corrected QT interval (QTc) during intravenous argatroban infusion in patients undergoing percutaneous coronary intervention (PCI).

Secondary objectives:

* Determination of the QTc interval after sufficient wash-out period by ECG-3 which needed to be performed > 8 but ≤ 28 hours after termination of prolonged argatroban infusion.
* Investigation of dependence of QTc interval on gender and applied doses.
* Determination of coagulation status during argatroban therapy.
* Assessment of safety-related events within the scope of anticoagulation with argatroban, for example bleeding events or thromboembolic events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stable CAD or unstable angina (troponin negative, i.e. within the normal range for the study site) with low to moderate anatomic risk.
* Patient required elective percutaneous coronary angioplasty or stent insertion with an approved device in one or more de novo-treated or re-stenotic lesions in native vessels.
* Patient was on adequate platelet inhibition therapy after having received a loading dose with ASA and clopidogrel before start of intervention (this additional inclusion criterion was introduced with study protocol version 1.6, dated 14.12.2018)
* Willingness to give written informed consent, written consent for data protection (legal requirement in Germany "datenschutzrechtliche Einwilligung") and willingness to participate and to comply with the requirements of the study protocol.
* The patient (female/male) was at least 18 years of age.
* Baseline ECG without changes that impair assessment of QTc interval.

Exclusion Criteria:

* Patient was indicated for highly complex 3-vessel intervention.
* The female patient was pregnant (exclusion by routine urine test) or was nursing during therapy period.
* Patients who were currently participating in another clinical trial or patients who participated in another clinical trial during the last 3 months prior to study start (date of treatment visit).
* History of drug, alcohol or chemical abuse within 6 months prior to study start.
* Planned surgical intervention other than study procedure within 7 days after study start.
* Any condition, which contraindicated the use of argatroban, or endangered the patient if he/she participated in this study.

Factors influencing QTc interval:

* Marked baseline prolongation of QTc interval (repeated demonstration of a QTc interval > 450 ms at baseline ECG).
* A history of risk factors of Torsade de pointes (e.g. heart failure, hypokalemia, family history of Long QT Syndrome).
* Known intraventricular conduction disturbance.
* Bradycardia: heart rate < 45 min-1.
* Electrolyte level outside normal range (according to laboratory's reference values).
* The use of concomitant medications that interfered with the QTc interval.
* Intake of digitalis within the last 2 weeks before study start.
* Acute myocardial infarction or troponin-positive unstable angina.

Factors inhibiting use of argatroban in this study:

* Intolerance to ingredients of Argatra® (sorbitol).
* Known cirrhosis, hepatitis, clinically significant hepatic disorder at study start and/or history of clinically relevant hepatic disorder.
* Current hepatic disorder indicated by laboratory liver profile at screening: Bilirubin, AST/SGOT, ALT/SGPT, gammaGT > 3.0 times upper limit of the normal (ULN).
* Renal insufficiency indicated by laboratory renal profile at study start: GFR < 35 ml/min.
* Uncontrolled hypertension (defined as blood pressure >180/120 mmHg).
* If any form of heparin was taken prior to study start and aPTT ≥ 35 s.
* Intake of direct oral anticoagulants (DOAC) within 1 month prior to study start.
* If anticoagulants of type of vitamin K antagonists (VKA) were taken prior to study start and INR >1.2.
* Platelet count <125 x 109/l.
* Documented coagulation disorder or bleeding diathesis.
* Uncontrolled haemorrhage within the past 3 months.
* Uncontrolled peptic ulcer disease or gastrointestinal bleeding within the past 3 months.
* Cerebral aneurysm.
* Haemorrhagic stroke or ischaemic stroke in the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deputy General Manager Scientific Medical Affairs, Study Director — Tanabe Pharma GmbH
Locations (2):
- Germany (2):
  - University Hospital Frankfurt, Frankfurt am Main, Hesse
  - Herz-Kreislauf-Zentrum Klinikum Hersfeld-Rotenburg, Rotenburg an der Fulda, Hesse

RESULTS

PARTICIPANT FLOW:
Groups:
- Argatroban Intravenous (i.v.) Bolus & i.v. Infusion: i.v. bolus of 300 μg/kg argatroban administered over a span of 3 to 5 minutes followed by the i.v. infusion of argatroban at 20 μg/kg/min until the end of the procedure.
Period: Overall Study
Arm/Group | Argatroban Intravenous (i.v.) Bolus & i.v. Infusion
Started | 50
Completed | 49
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Argatroban Intravenous (i.v.) Bolus & i.v. Infusion
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 49
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in QTc Interval Between ECG-2 and ECG-1 (ITT Population)
Description: It was investigated if a mean QTc prolongation of more than 10 ms occurred between ECG-2 and ECG-1
Time Frame: ECG-2 was recorded immediately after cardiac intervention when patient was fully anticoagulated with argatroban and ECG-1 was recorded at baseline prior to first bolus dose of argatroban (argatroban-free status).
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Argatroban Intravenous (i.v.) Bolus & i.v. Infusion (ITT Population): i.v. bolus of 300 μg/kg argatroban administered over a span of 3 to 5 minutes followed by the i.v. infusion of argatroban at 20 μg/kg/min until the end of the procedure.
Arm/Group | Argatroban Intravenous (i.v.) Bolus & i.v. Infusion (ITT Population)
Number analyzed (Participants) | 50
milliseconds | 0.94 (46.37)

2. Primary Outcome: Mean Difference in QTc Interval Between ECG-2 and ECG-1 (ITT Population/Subgroup Male or Female)
Description: It was investigated if a mean QTc prolongation of more than 10 ms occurred between ECG-2 and ECG-1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Argatroban Intravenous (i.v.) Bolus & i.v. Infusion (ITT Population/Sub Group Male): i.v. bolus of 300 μg/kg argatroban administered over a span of 3 to 5 minutes followed by the i.v. infusion of argatroban at 20 μg/kg/min until the end of the procedure in Subgroup Male.
- Argatroban Intravenous (i.v.) Bolus & i.v. Infusion (ITT Population/Sub Group Female): i.v. bolus of 300 μg/kg argatroban administered over a span of 3 to 5 minutes followed by the i.v. infusion of argatroban at 20 μg/kg/min until the end of the procedure in Subgroup Female.
Arm/Group | Argatroban Intravenous (i.v.) Bolus & i.v. Infusion (ITT Population/Sub Group Male) | Argatroban Intravenous (i.v.) Bolus & i.v. Infusion (ITT Population/Sub Group Female)
Number analyzed (Participants) | 39 | 11
milliseconds | -5.8936 (46.4072) | 25.1460 (39.0616)

3. Primary Outcome: Mean Difference in QTc Interval Between ECG-2 and ECG-1 (ITT Population/Centre 01 or Centre 02)
Description: It was investigated if a mean QTc prolongation of more than 10 ms occurred between ECG-2 and ECG-1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Argatroban Intravenous (i.v.) Bolus & i.v. Infusion (ITT Population/Centre 01): i.v. bolus of 300 μg/kg argatroban administered over a span of 3 to 5 minutes followed by the i.v. infusion of argatroban at 20 μg/kg/min until the end of the procedure in Centre 01.
- Argatroban Intravenous (i.v.) Bolus & i.v. Infusion (ITT Population/Centre 02): i.v. bolus of 300 μg/kg argatroban administered over a span of 3 to 5 minutes followed by the i.v. infusion of argatroban at 20 μg/kg/min until the end of the procedure in Centre 02.
Arm/Group | Argatroban Intravenous (i.v.) Bolus & i.v. Infusion (ITT Population/Centre 01) | Argatroban Intravenous (i.v.) Bolus & i.v. Infusion (ITT Population/Centre 02)
Number analyzed (Participants) | 25 | 25
milliseconds | 15.0046 (44.9538) | -13.1343 (44.2363)

4. Secondary Outcome: Proportion of Patients With a Prolongation of QTc Interval to >500 ms at ECG-2
Description: Number of patients of ITT population exhibiting QTc interval of > 500 ms
Time Frame: ECG-2 immediately after argatroban infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Argatroban Intravenous (i.v.) Bolus & i.v. Infusion
Number analyzed (Participants) | 50
Participants | 1

ADVERSE EVENTS:
Time Frame: i.v. bolus of 300 μg/kg argatroban administered over a span of 3 to 5 minutes followed by the i.v. infusion of argatroban at 20 μg/kg/min until the end of the procedure.
Description: All AEs encountered during the clinical study will be reported on the AE page of the CRF.
Arm/Group | Argatroban Intravenous (i.v.) Bolus & i.v. Infusion
All-Cause Mortality (participants affected / at risk) | 1/50
Serious Adverse Events (participants affected / at risk) | 3/50
Other Adverse Events (participants affected / at risk) | 4/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Argatroban Intravenous (i.v.) Bolus & i.v. Infusion (N=50)
Vascular stent thrombosis (Vascular disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 3
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Argatroban Intravenous (i.v.) Bolus & i.v. Infusion (N=50)
Electrocardiogram ST segment depression (Investigations) | 1
Sinus bradycardia (Cardiac disorders) | 1
Hypertension (Blood and lymphatic system disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT05740371/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT05740371/SAP_001.pdf